CLINICAL TRIAL: NCT03213275
Title: The Premature Gut Microbiome and the Influence on Neonatal Immunity, Brain Development and White Matter Injury
Acronym: PreMiBraIn
Status: Active, not recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: University of Vienna (Other)
Responsible Party: Principal Investigator, Lukas Wisgrill, Dr., Medical University of Vienna
Other Study IDs: PreMiBraIn
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Microbiome; Neurodevelopment Outcome; Immunology
Keywords: Extremely premature infants; gut-immune-brain axis; neonatal brain injury; gut microbiome; neurodevelopmental outcome; neonatal immunity
MeSH Terms: interventions — Immunologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Microbiome Sequencing, Neurophysiologic Assessment, Immunological test — Stool sampling, aEEG, VEP, NIRS, ydTCR, Treg, biomarker

SUMMARY:
Recent advances in neonatal intensive care have dramatically increased the survival rate of extremely premature infants but the number of survivors with severe morbidity and lifelong neurodevelopmental impairment remains high. Perinatal white matter injury is the predominant form of brain injury in premature infants, often leading to adverse neurodevelopmental outcome. Intrauterine and neonatal infection and inflammation have been identified as major risk factors of neonatal brain injury. The fragile gut microbiome of premature infants seems to play an important role in health and disease as distortions of the microbiome occur prior to sepsis and necrotizing enterocolitis. Furthermore, the close link of the gut microbiome to neurological and psychiatric diseases in animal models suggests that the microbiome may influence brain maturation and development in preterm infants. Recent studies have underlined the importance of regulatory T cells as well as γδ T cells in brain injury, which can be directly influenced by the gut microbiome. It is therefore likely that an underdeveloped or distorted gut microbiome affects host immune response and may be a risk factor for neurodevelopmental disabilities in extremely premature infants who are already challenged by the unphysiologic early extrauterine environment after premature birth which affects maturation of the gut microbiome and immune system as well as neurophysiological maturation alike.

Therefore, the overarching aim of the PreMiBraIn study is to elucidate the role of the gut-immune-brain axis on neonatal brain injury and its impact on long-term neurodevelopmental outcome of extremely premature infants. The study cohort will consist of a total of 60 extremely premature infants with a gestational age < 28 weeks and birth weight < 1000 grams. The investigators seek to characterize the orchestrated dynamics of the maturation of the gut microbiome and the subsequent impact on maturation of innate and adaptive immune mechanisms as well as neurophysiological maturation and neurodevelopmental outcome. Furthermore, the investigators will assess the value of the microbiome as a prognostic indicator for neonatal brain injury as well as short- and long-term neurodevelopmental outcome of extremely premature infants.

This goal will be achieved by state-of-the-art techniques using 16s rRNA gene sequencing of the gut microbiome, holistic analysis of T cell biology using flow cytometry, whole transcriptome analysis and proteomics as well as neurophysiological measurements (amplitude-integrated EEG, near-infrared spectroscopy, visual evoked potentials) and cranial MRI of extremely premature infants. Short- and long-term neurological outcome will be investigated using Bayley Scales of Infant Development, Third Edition at one and two years corrected age, and Kaufmann-Assessment Battery for Children at five years of age. The investigators expect to find microbiome signatures that are predictive for later neurodevelopmental disabilities which may then be used for early screening and intervention and may suggest personalized therapeutic options. The prospects of precision medicine targeting the gut-immune-brain axis in extremely premature infants hold the opportunity to improve the overall outcome of these high-risk patients.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age < 28+0 weeks
* Birth weight < 1000 gram

Exclusion Criteria:

* chromosomal aberrations
* congenital malformations
* inborn metabolic disorders
* maternal chronic infectious diseases
* missing informed consent

Max Age: 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Extreme premature infants
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2025-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Neurodevelopmental outcome with corrected age of two and five years | Eight Years

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Wisgrill, M.D., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria